CLINICAL TRIAL: NCT00335998
Title: Phase I Study of Intravenous Triapine® (IND #68338) in Combination With Pelvic Radiation Therapy With or Without Weekly Intravenous Cisplatin Chemotherapy for Locally Advanced Cervical, Vaginal, or Pelvic Gynecologic Malignancies.
Brief Title: Phase I Study of Intravenous Triapine (IND # 68338) in Combination With Pelvic Radiation Therapy With or Without Weekly Intravenous Cisplatin Chemotherapy for Locally Advanced Cervical, Vaginal, or Pelvic Gynecologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03126; CASE 1805; U01CA062502 (NIH)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Cervical Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Vaginal Cancer; Recurrent Vulvar Cancer; Stage III Vaginal Cancer; Stage IIIA Cervical Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Vulvar Cancer; Stage IIIB Cervical Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Vulvar Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Vulvar Cancer; Stage IV Ovarian Epithelial Cancer; Stage IVA Cervical Cancer; Stage IVA Vaginal Cancer; Stage IVB Cervical Cancer; Stage IVB Vaginal Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma, Ovarian Epithelial; Vaginal Neoplasms; Vulvar Neoplasms | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; Brachytherapy; Therapeutics; Cisplatin

ARMS (1):
- Treatment (triapine) (Experimental): Group 1: Patients undergo external-beam pelvic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients also receive 3-AP IV over 2 hours on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33 and cisplatin IV over 1½ hours on day 2, 9, 16, 23, and 30.
  Group 2: Patients undergo external-beam pelvic radiotherapy and receive 3-AP as in group 1.
  In both groups, patients undergo intracavitary or interstitial brachytherapy at least once weekly for 3-5 weeks during or after external-beam radiotherapy as per standard of care.
  Interventions: Drug: triapine; Other: laboratory biomarker analysis; Radiation: external beam radiation therapy; Radiation: brachytherapy; Drug: cisplatin; Other: pharmacological study

INTERVENTIONS:
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Other: laboratory biomarker analysis — Correlative studies
Radiation: external beam radiation therapy — Undergo external beam radiation therapy
  Other Names: EBRT
Radiation: brachytherapy — Undergo intracavitary or interstitial brachytherapy
  Other Names: low-LET implant therapy; radiation brachytherapy; therapy, low-LET implant
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy, such as 3-AP and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. 3-AP may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. 3-AP and cisplatin may make tumor cells more sensitive to radiation therapy. Giving 3-AP and external-beam radiation therapy together with cisplatin may kill more tumor cells. This phase I trial is studying the side effects and best dose of 3-AP when given together with external-beam radiation therapy with or without cisplatin in treating patients with gynecologic cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of Triapine® when given in combination with pelvic radiotherapy with or without weekly intravenous cisplatin chemotherapy.

II. To determine the dose limiting toxicity (DLT) of Triapine® when given in combination with pelvic radiotherapy with or without weekly intravenous cisplatin chemotherapy.

III. To determine the safety and sequelae of intravenous Triapine® when given in combination with pelvic radiotherapy with or without weekly intravenous cisplatin chemotherapy.

SECONDARY OBJECTIVES:

I. Evaluation of intravenous Triapine®'s targeted inhibition of ribonucleotide reductase through tumor tissue biopsy at pretreatment evaluation and during external beam radiotherapy (Day 10).

II. Serial monitoring of methemoglobin levels during therapy given Triapine®'s iron chelating properties.

OUTLINE: This is a multicenter, dose-escalation study of 3-AP. Patients are assigned to 1 of 2 treatment groups based on eligibility* to receive cisplatin (yes vs no).

NOTE: *Patients who refuse or are not candidates for cisplatin chemotherapy due to prior platinum adverse sensitivity, active neuropathy, or comobid illness, as determined by the treating physician, are eligible to receive 3-AP alone with pelvic radiotherapy.

Group 1: Patients undergo external-beam pelvic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients also receive 3-AP IV over 2 hours on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33 and cisplatin IV over 1½ hours on day 2, 9, 16, 23, and 30.

Group 2: Patients undergo external-beam pelvic radiotherapy and receive 3-AP as in group 1.

In both groups, patients undergo intracavitary or interstitial brachytherapy at least once weekly for 3-5 weeks during or after external-beam radiotherapy as per standard of care.

Cohorts of 3-6 patients in group 1 and 1-3 patients in group 2 receive escalating doses of 3-AP until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Patients undergo blood draws on days 1 and 10 before treatment with 3-AP and at 2, 4, 6, and 24 hours after starting treatment to assess methemoglobin levels and 3-AP plasma levels. Patients also undergo punch biopsy on days 1 and 10 to determine R2 protein levels by Western blot analysis, ribonucleotide reductase R2 protein levels by flow cytometry, and cytidine deoxyphosphate reductase assay.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically-proven primary or recurrent locally advanced cervical, vaginal, or vulvar cancers not amenable to curative surgical resection alone are eligible
* Patients with pathologically-proven recurrent or persistent epithelial ovarian or endometrial cancer a) not amenable to curative surgical resection alone, b) are planned for pelvic radiotherapy, and c) are amenable to tumor biopsy through the vaginal canal are eligible
* Patients with other active invasive malignancies are excluded; patients with prior malignancies in remission for at least six months and not being currently treated are eligible; patients are excluded if their previous cancer treatment as determined by their treating physicians contraindicates this protocol therapy or if they have received prior low abdominal or pelvic radiotherapy that would contribute radiation dose that would exceed tolerance of normal tissues (as determined by the principal investigator or co-investigators); for patients relapsing at least four weeks after initial surgery or chemotherapy, they must have fully recovered from side effects of prior treatment, have measurable disease in the pelvis; measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques (CT, MRI, x-ray or as >= 10 mm with spiral CT scan; patients with metastatic disease to extra-pelvic sites are eligible if pelvic radiotherapy is planned as primary management of the site of pelvic disease. There is no numerical limit on prior chemotherapy regimens previously received
* ECOG performance status 0-2; (Karnofsky >= 50%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 2.0 mg/dL
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* PT/aPTT =< 1.5 X institutional upper limit of normal
* Patients should have a serum creatinine =< 1.5mg/dL to receive weekly intravenous cisplatin chemotherapy; patients whose serum creatinine is between 1.5 and 1.9 mg/dL are eligible for cisplatin chemotherapy if the estimated creatinine clearance is >= 30 ml/min; for the purpose of estimating the creatinine clearance, the formula of Jelliffe should be used: CCr = 0.9{98-[0.8(age-20)]}/Scr where CCr is the estimated creatinine clearance, age is patient's age in years (from 20-80), and Scr is the serum creatinine in mg/dL; patients eligible for cisplatin chemotherapy will also receive intravenous Triapine®; patients who have refused or are not candidates for cisplatin chemotherapy as defined above, have prior platinum adverse sensitivity, have active neuropathy, or have intercurrent co-morbid illness as determined by treating physicians will receive intravenous Triapine® alone with pelvic radiation; to receive Triapine® alone with pelvic radiotherapy, patients must have a serum creatinine =< 2.0mg/dL
* The effects of Triapine® on the developing human fetus are unknown; for this reason and because heterocyclic carboxaldehyde thiosemicarbazones as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of Triapine® will be determined following review of their case by the Principal Investigator
* Ability to undergo and the willingness to sign a written informed consent for placement of a PICC line or a central venous catheter
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are excluded
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Triapine® or other agents used in study
* Patients unable to receive intravenous chemotherapies as a consequence of poor vascular access (for example, patient receiving hemodialysis) are ineligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, known inadequately controlled hypertension, significant pulmonary disease including dyspnea at rest, patients requiring supplemental oxygen, or poor pulmonary reserve; proteinuria or clinically significant renal function impairment (baseline serum creatinine > 2mg/dL), or psychiatric illness/social situations that would limit compliance with study requirements are excluded
* Patients with known glucose-6-phosphate dehydrogenase deficiency (G6PD) are excluded
* Pregnant women are excluded from this study because Triapine® is a heterocyclic carboxaldehyde thiosemicarbazone with the potential for teratogenic or abortifacient effects; screening b-hcg levels and diagnostic tests will be used to determine eligibility; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Triapine®, breastfeeding should be discontinued if the mother is treated with Triapine®; these potential risks may also apply to other agents used in this study
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Triapine®; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-03; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Toxicity of radiotherapy and Triapine® combination therapy as documented by dose-limiting toxicities (DLTs) using Common Terminology Criteria for Adverse Events (CTCAE) criteria, version 3.0 | Up to 12 weeks
MTD of Triapine® when given in combination with pelvic radiotherapy with or without weekly intravenous cisplatin chemotherapy | 12 weeks

SECONDARY OUTCOMES:
RR R2 enzyme quantity | Baseline
  Paired T-tests will be used to compare RR R2 enzyme quantity and activity before and after treatment. %MHgb levels will be tracked over time with corresponding pharmacokinetic and biopsy analyses and tested for time course correlations with plasma Triapine® concentrations.
RR R2 enzyme quantity | Day 10
  Paired T-tests will be used to compare RR R2 enzyme quantity and activity before and after treatment. %MHgb levels will be tracked over time with corresponding pharmacokinetic and biopsy analyses and tested for time course correlations with plasma Triapine® concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kunos, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States